CLINICAL TRIAL: NCT04199572
Title: Synergistic Effect Of Parenteral Diclofenac And Paracetamol In The Pain Management Of Acute Limb Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Isma Qureshi, Academic Research Associate, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRGC-04-NI-17-099
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Musculoskeletal Injury
MeSH Terms: interventions — Diclofenac; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Combination 1- Diclofenac Placebo Paracetamol (Oral) Combination 2- Diclofenac Paracetamol (IV) Placebo Combination 3- Diclofenac Placebo Placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The physicians, participants, nurses and the outcome assessor will all be blinded to the intervention. The trial packets will be prepared containing the active drugs and placebos.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diclofenac and Oral Paracetamol (Experimental): Diclofenac (75mg intramuscular), Placebo (100ml intravenous Normal Saline), Paracetamol (per oral 1gm)
  Interventions: Drug: Diclofenac and Paracetamol
- Diclofenac and IV Paracetamol (Experimental): Diclofenac (75mg intramuscular), Paracetamol (intravenous1gm in 100ml solution), Placebo (sugar tablets)
  Interventions: Drug: Diclofenac and Paracetamol
- Diclofenac and Placebo (Experimental): Diclofenac (75mg intramuscular),Placebo (100ml intravenous Normal Saline),Placebo (sugar tablets)
  Interventions: Drug: Diclofenac and Paracetamol

INTERVENTIONS:
Drug: Diclofenac and Paracetamol — analgesic effect of diclofenac along with either Oral versus Intravenous paracetamol versus placebo
  Other Names: Placebo

SUMMARY:
Acute limb injury is a common reason to visit an emergency department worldwide. Intense pain related to the injury is always a concern for an emergency physician and requires effective analgesia within the shortest possible time. Non-steroidal anti-inflammatory drugs (NSAIDs), opioids and paracetamol are the commonly used drugs in an emergency department. The choice of analgesia should be established by its efficacy, logistics involved and route of administration. There is good evidence about NSAIDs being the first line analgesia and paracetamol is reported to have the narcotic sparing effect, either alone or as an adjunctive treatment in different settings. The synergistic effect of paracetamol with diclofenac in acute limb injuries related pain management lacks good- quality evidence. Therefore investigators proposed a large, well designed, randomized double-blind trial to develop high-quality evidence. The study aims to assess the efficacy of paracetamol in addition to diclofenac, and compare the difference between oral and intravenous paracetamol administration in acute limb injuries in the emergency department.

DETAILED DESCRIPTION:
Injuries account for a large burden of mortality and morbidity in the state of Qatar and worldwide. Among all the acute injuries, limb injuries are very common. Immense pain of patients on presentation is the matter of concern and requires effective analgesia within the shortest possible time.

Most patients with acute limb injuries are treated with, the commonly used analgesics like non-steroidal anti-inflammatory drugs (NSAIDs), opioids, and paracetamol in the ED. The choice of analgesic should be established by its efficacy, logistics involved, and route of drug administration. Few studies reported that intravenous route is more effective than the intramuscular route, due to its faster absorption and ease of titration. In many ED's intramuscular injectable drugs like NSAIDs are commonly used. Being, readily available and technically faster to administer. There is concern about the use of IM diclofenac in some countries because of possible intramuscular complications; however, most are reported cases in a small proportion (<2 per million doses used). Oral medications are also very commonly used and usually self-administered by the patients with duration of onset being in minutes to an hour. There is good evidence about NSAIDs being the first line analgesic in the management of acute painful conditions such as renal colic. Intramuscular diclofenac is shown to provide safe, effective, and sustained pain relief in addition to being logistically easier to administer. Paracetamol being a centrally acting inhibitor of cyclooxygenases has been reported safe alternative to opioids and equally effective analgesic in the ED with fewer side effects and contraindications. In addition, paracetamol is reported to have the narcotic sparing effect, either alone or as an adjunctive treatment in different settings including post-op pain, cancer pain, and regional anesthesia. The synergistic effect of paracetamol with diclofenac in acute limb injury related- pain management lacks good-quality evidence.

Hamad General Hospital Emergency Department (HGH-ED) is the major emergency department (ED) in Doha; Qatar; and offers tertiary level care for emergency conditions. It is also one of the busiest ED's in the world with an annual patient attendance of 0.5 million. Patients with acute limb injuries account for about 25% of the total ED visits. At HGH-ED, intramuscular diclofenac is the analgesia of choice for the management of acute pain of moderate to severe intensity. However, 40-50% of these patients require additional analgesia in the form of opioids or paracetamol. The efficacy of combined analgesia approach, and the difference by route of drug administration in acute ED pain management is yet to be assessed. Therefore investigators proposed a large, well designed, randomized, double- blind trial to develop high-quality evidence. This study aims to assess the efficacy of paracetamol in addition to diclofenac, and compare the difference between oral and intravenous paracetamol administration in acute limb injury pain management in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years upto 65 years
* Vitals Stable
* musculoskeletal limb injury
* initial pain score of 5 or more on a NRS (numerical rating scale)

Exclusion Criteria:

* Patient received any pain medication prior to 8 hours
* Allergies to either diclofenac or paracetamol
* Contraindication to the study drugs
* CVA
* Bronchial asthma
* GI bleeding
* Renal impairment
* Asthma
* Pregnancy and nursing
* Unstable traumatic patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
To compare the difference in mean pain reduction amongst the three groups: numerical rating scale | 30 minutes
  Pain score on a numerical rating scale (NRS). The scale is a 11 point scale where 0 is no pain and 10 is the worst pain ever.

SECONDARY OUTCOMES:
To compare the difference in proportion of patients achieving 50% or more pain relief amongst the three groups | 30 minutes
  Pain score on a numerical rating scale (NRS). The scale is a 11 point scale where 0 is no pain and 10 is the worst pain ever.
Requirement of rescue analgesia in each group of participants | 30 minutes
  Pain score on a numerical rating scale (NRS). The scale is a 11 point scale where 0 is no pain and 10 is the worst pain ever.
The adverse event rate in three groups | 90 minutes
  any adverse event recorded
Time to analgesia effect, to achieve 50% reduction, and to NRS <=2 | 90 minutes
  Pain score on a numerical rating scale (NRS). The scale is a 11 point scale where 0 is no pain and 10 is the worst pain ever.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tramer MR, Williams JE, Carroll D, Wiffen PJ, Moore RA, McQuay HJ. Comparing analgesic efficacy of non-steroidal anti-inflammatory drugs given by different routes in acute and chronic pain: a qualitative systematic review. Acta Anaesthesiol Scand. 1998 Jan;42(1):71-9. doi: 10.1111/j.1399-6576.1998.tb05083.x. PMID 9527748
- [Background] Khalili G, Janghorbani M, Saryazdi H, Emaminejad A. Effect of preemptive and preventive acetaminophen on postoperative pain score: a randomized, double-blind trial of patients undergoing lower extremity surgery. J Clin Anesth. 2013 May;25(3):188-92. doi: 10.1016/j.jclinane.2012.09.004. Epub 2013 Apr 6. PMID 23567482
- [Result] Aarons L, Ogungbenro K. Optimal design of pharmacokinetic studies. Basic Clin Pharmacol Toxicol. 2010 Mar;106(3):250-5. doi: 10.1111/j.1742-7843.2009.00533.x. Epub 2010 Jan 20. PMID 20102362
- [Result] Krug EG, Sharma GK, Lozano R. The global burden of injuries. Am J Public Health. 2000 Apr;90(4):523-6. doi: 10.2105/ajph.90.4.523. PMID 10754963
- [Result] Macintyre PE, Schug SA, Scott DA. Acute pain management: the evidence grows. Med J Aust. 2006 Feb 6;184(3):101-2. doi: 10.5694/j.1326-5377.2006.tb00144.x. PMID 16460291
- [Result] Tveita T, Thoner J, Klepstad P, Dale O, Jystad A, Borchgrevink PC. A controlled comparison between single doses of intravenous and intramuscular morphine with respect to analgesic effects and patient safety. Acta Anaesthesiol Scand. 2008 Aug;52(7):920-5. doi: 10.1111/j.1399-6576.2008.01608.x. PMID 18702754
- [Result] Tuomilehto H, Kokki H. Parenteral ketoprofen for pain management after adenoidectomy: comparison of intravenous and intramuscular routes of administration. Acta Anaesthesiol Scand. 2002 Feb;46(2):184-9. doi: 10.1034/j.1399-6576.2002.460211.x. PMID 11942868
- [Result] Hindle A, Spedding R. Managing acute renal colic. Intramuscular diclofenac should be avoided. BMJ. 2003 Mar 1;326(7387):502. doi: 10.1136/bmj.326.7387.502. No abstract available. PMID 12609956
- [Result] Wright PJ, English PJ, Hungin AP, Marsden SN. Managing acute renal colic across the primary-secondary care interface: a pathway of care based on evidence and consensus. BMJ. 2002 Dec 14;325(7377):1408-12. doi: 10.1136/bmj.325.7377.1408. No abstract available. PMID 12480861
- [Result] Moran CP, Courtney AE. Managing acute and chronic renal stone disease. Practitioner. 2016 Feb;260(1790):17-20, 2-3. PMID 27032222
- [Result] Pathan SA, Mitra B, Straney LD, Afzal MS, Anjum S, Shukla D, Morley K, Al Hilli SA, Al Rumaihi K, Thomas SH, Cameron PA. Delivering safe and effective analgesia for management of renal colic in the emergency department: a double-blind, multigroup, randomised controlled trial. Lancet. 2016 May 14;387(10032):1999-2007. doi: 10.1016/S0140-6736(16)00652-8. Epub 2016 Mar 16. PMID 26993881
- [Result] Babl FE, Theophilos T, Palmer GM. Is there a role for intravenous acetaminophen in pediatric emergency departments? Pediatr Emerg Care. 2011 Jun;27(6):496-9. doi: 10.1097/PEC.0b013e31821d8629. PMID 21629146
- [Result] Serinken M, Eken C, Turkcuer I, Elicabuk H, Uyanik E, Schultz CH. Intravenous paracetamol versus morphine for renal colic in the emergency department: a randomised double-blind controlled trial. Emerg Med J. 2012 Nov;29(11):902-5. doi: 10.1136/emermed-2011-200165. Epub 2011 Dec 20. PMID 22186009
- [Result] Craig M, Jeavons R, Probert J, Benger J. Randomised comparison of intravenous paracetamol and intravenous morphine for acute traumatic limb pain in the emergency department. Emerg Med J. 2012 Jan;29(1):37-9. doi: 10.1136/emj.2010.104687. Epub 2011 Mar 1. PMID 21362724
- [Result] Bektas F, Eken C, Karadeniz O, Goksu E, Cubuk M, Cete Y. Intravenous paracetamol or morphine for the treatment of renal colic: a randomized, placebo-controlled trial. Ann Emerg Med. 2009 Oct;54(4):568-74. doi: 10.1016/j.annemergmed.2009.06.501. Epub 2009 Jul 31. PMID 19647342
- [Result] Grissa MH, Claessens YE, Bouida W, Boubaker H, Boudhib L, Kerkeni W, Boukef R, Nouira S. Paracetamol vs piroxicam to relieve pain in renal colic. Results of a randomized controlled trial. Am J Emerg Med. 2011 Feb;29(2):203-6. doi: 10.1016/j.ajem.2009.09.019. Epub 2010 Oct 8. PMID 20934829
- [Result] Sinatra RS, Jahr JS, Reynolds LW, Viscusi ER, Groudine SB, Payen-Champenois C. Efficacy and safety of single and repeated administration of 1 gram intravenous acetaminophen injection (paracetamol) for pain management after major orthopedic surgery. Anesthesiology. 2005 Apr;102(4):822-31. doi: 10.1097/00000542-200504000-00019. PMID 15791113
- [Result] Olonisakin RP, Amanor-Boadu SD, Akinyemi AO. Morphine-sparing effect of intravenous paracetamol for post operative pain management following gynaecological surgery. Afr J Med Med Sci. 2012 Dec;41(4):429-36. PMID 23672109
- [Derived] Qureshi I, S Qureshi R, Harris T, A Pathan S, Malik AME, Babiker ME, Jamali MA, Bhutta ZA, Thomas SH. A Randomized Trial Evaluating the Synergistic Effect of Parenteral Diclofenac and Paracetamol for Pain Management in Adult Males With Acute Limb Injury. Pain Res Manag. 2026 Jan 31;2026:5587917. doi: 10.1155/prm/5587917. eCollection 2026. PMID 41623940